CLINICAL TRIAL: NCT04044794
Title: Daily Self-Weighing for Obesity Management in Primary Care
Acronym: SWOP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Indiana University (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK118939 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity
Keywords: weight management; body weight; behavioral; weighing
MeSH Terms: conditions — Overweight; Obesity; Body Weight; Behavior | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participants randomly assigned to this arm will receive standardized weight management educational materials plus a monetary gift of $60 that can be used to purchase health-promoting supplies to support weight management.
  Interventions: Behavioral: Standard Care
- Daily Self-Weighing (Experimental): Participants randomly assigned to this arm will receive standardized weight management educational materials plus a commercially available wireless scale. Participants will be instructed to weigh daily and view their weight on the scale's digital display.
  Interventions: Behavioral: Daily Self-Weighing

INTERVENTIONS:
Behavioral: Standard Care — Standard care includes standardized educational materials to promote self-management of body weight along with provision of $60 for participants to purchase supplies or equipment to facilitate weight management.
  Arms: Standard Care
Behavioral: Daily Self-Weighing — Participants will receive a wireless digital scale and will be asked to keep the scale in their home, weigh daily at the same time, and view their weight trajectory on the scale's digital display.
  Arms: Daily Self-Weighing

SUMMARY:
Many adults with obesity continue to gain weight even though they do not want to. This project will test the effects of a primary care intervention in which people with obesity receive an electronic scale and recommendations to weigh themselves daily. This will help us understand whether daily self-weighing might be a way to prevent continued weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-65 years
* Body mass index (BMI) 30 - 50 kg/m2
* Receives care at one of the participating primary care clinics
* Resides in one location at least 5 days each week
* Possesses a smartphone with data plan
* Wi-Fi or Bluetooth internet connection in home

Exclusion Criteria:

* Pregnancy or anticipating pregnancy during study duration. This is a weight loss study and weight gain/loss due to pregnancy and/or delivery would confound study results. Additionally, weight loss is not recommended for pregnant women.
* Unwilling or unable to do any of the following: give informed consent, accept random assignment, attend five measurement assessments
* Likely to relocate and no longer be seen at UAB primary care in the next 2 years
* Weight loss ≥5% of body weight in past 6 months (other than postpartum)
* Weight >180 kg (396lbs) due to the limitation of the scale being used.
* Current participation in another weight loss study
* Bariatric surgery or revision in the past two years
* Prescription weight loss medications within the past 6 months
* Another household member already participating in the study
* Potential participants living farther than 50 miles driving distance from UAB will be excluded from the study. It is expected that those living farther away will be more difficult to retain as study participants.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline to month 6 | 6 months
  Body weight measured to the nearest 0.1 kg using a calibrated electronic scale
Change in body weight from baseline to month 12 | 12 months
  Body weight measured to the nearest 0.1 kg using a calibrated electronic scale
Change in body weight from baseline to month 18 | 18 months
  Body weight measured to the nearest 0.1 kg using a calibrated electronic scale
Change in body weight from baseline to month 24 | 24 months
  Body weight measured to the nearest 0.1 kg using a calibrated electronic scale

SECONDARY OUTCOMES:
Average number of weight control behaviors endorsed on the Weight Control Practices Survey at month 6 | baseline to month 6
  A modified version of the 23-item Weight Control Practices Survey will assess a variety of strategies for weight control, including participation in structured programs and/or self-directed weight control behaviors (e.g., reducing fat intake, maintaining food records, increasing physical activity, frequency of self-weighing). The survey measures presence and duration (in weeks) of each behavior.
Average number of weight control behaviors endorsed on the Weight Control Practices Survey at month 12 | month 6 to month 12
  A modified version of the 23-item Weight Control Practices Survey will assess a variety of strategies for weight control, including participation in structured programs and/or self-directed weight control behaviors (e.g., reducing fat intake, maintaining food records, increasing physical activity, frequency of self-weighing). The survey measures presence and duration (in weeks) of each behavior.
Average number of weight control behaviors endorsed on the Weight Control Practices Survey at month 18 | month 12 to month 18
  A modified version of the 23-item Weight Control Practices Survey will assess a variety of strategies for weight control, including participation in structured programs and/or self-directed weight control behaviors (e.g., reducing fat intake, maintaining food records, increasing physical activity, frequency of self-weighing). The survey measures presence and duration (in weeks) of each behavior.
Average number of weight control behaviors endorsed on the Weight Control Practices Survey at month 24 | month 18 to month 24
  A modified version of the 23-item Weight Control Practices Survey will assess a variety of strategies for weight control, including participation in structured programs and/or self-directed weight control behaviors (e.g., reducing fat intake, maintaining food records, increasing physical activity, frequency of self-weighing). The survey measures presence and duration (in weeks) of each behavior.

OTHER OUTCOMES:
Mean self-efficacy score assessed by the Self-Efficacy for Weight Loss Trials Scale at month 12 | month 12
  Self-efficacy (i.e., confidence in one's ability to execute the behaviors required to meet a goal) for healthy eating, physical activity, and weight loss will be assessed with the 12-item Self-Efficacy for Weight Loss Trials Scale
Mean self-efficacy score assessed by the Self-Efficacy for Weight Loss Trials Scale at month 24 | month 24
  Self-efficacy (i.e., confidence in one's ability to execute the behaviors required to meet a goal) for healthy eating, physical activity, and weight loss will be assessed with the 12-item Self-Efficacy for Weight Loss Trials Scale
Mean score on the Eating Disorder Diagnostic Screening form at month 12 | month 12
  The 22-item Eating Disorder Diagnostic Screening will monitor symptoms of eating disorders
Mean score on the Eating Disorder Diagnostic Screening form at month 24 | month 24
  The 22-item Eating Disorder Diagnostic Screening will monitor symptoms of eating disorders
Mean score on the Body Shape Questionnaire-16A at month 12 | month 12
  The 16-item Body Shape Questionnaire-16A will monitor symptoms of body image disturbance
Mean score on the Body Shape Questionnaire-16A at month 24 | month 24
  The 16-item Body Shape Questionnaire-16A will monitor symptoms of body image disturbance
Mean score on the Patient Health Questionnaire-8 (PHQ-8) at month 12 | month 12
  The Patient Health Questionnaire-8 (PHQ-8) will monitor depressive symptoms
Mean score on the Patient Health Questionnaire-8 (PHQ-8) at month 24 | month 24
  The Patient Health Questionnaire-8 (PHQ-8) will monitor depressive symptoms
Healthcare utilization at month 12 assessed by the EuroQOL (EQ-5D-5L) | baseline to month 12
  Self-reported use of health care services (hospitalizations, ER/physician office visits, prescription drugs, etc.) and associated costs will be collected using the EuroQOL (EQ-5D-5L)
Healthcare utilization at month 24 assessed by the EuroQOL (EQ-5D-5L) | month 12 to month 24
  Self-reported use of health care services (hospitalizations, ER/physician office visits, prescription drugs, etc.) and associated costs will be collected using the EuroQOL (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will ensure all publications that result from project-related data will comply with the NIH public access policy and develop a system by which study data may be shared with other investigators within the scientific community. With UAB IRB permission, PI may develop a de-identified database, codebook, and mechanism by which data can be shared with qualified individuals/organizations. PI will keep a record of all individuals/res. teams who request/receive a copy of the data. Interested investigators will be asked to complete a request form stating specific aims of the analyses, analytic plan, available resources, proposed timeline, and goals. PI and team will review these requests to determine whether proposed analyses constitute significant exploration of the data, team has resources to complete request, and data will be adequately protected and managed. If any issues are problematic, PI and team will attempt to negotiate a fair resolution with investigators and NIH staff.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Dutton GR, Kinsey AW, Howell CR, Pisu M, Dobelstein AE, Allison DB, Xun P, Levitsky DA, Fontaine K. The daily Self-Weighing for Obesity Management in Primary Care Study: Rationale, design and methodology. Contemp Clin Trials. 2021 Aug;107:106463. doi: 10.1016/j.cct.2021.106463. Epub 2021 May 31. PMID 34082075